CLINICAL TRIAL: NCT06048185
Title: Long Term Follow-up for Participants Who Previously Received a Single Intravitreal Injection of MCO-010 Optogenetic Therapy in the STARLIGHT Study
Brief Title: Non-interventional Long Term Follow-up Study of Participants Previously Enrolled in the STARLIGHT Study
Acronym: SUSTAIN
Status: Active, not recruiting | Type: Observational
Sponsor: Nanoscope Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NTXLTFU-007
Record Dates: First submitted 2023-09-11; First posted 2023-09-21 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Stargardt Disease
Keywords: Eye Diseases; Retinal Degeneration; Retinal Dystrophy; Eye Diseases, Hereditary
MeSH Terms: conditions — Stargardt Disease; Eye Diseases; Retinal Degeneration; Retinal Dystrophies; Eye Diseases, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Biological: Gene Therapy Product-MCO-010 — The MCO-010 is an adeno-associated virus serotype 2-based vector carried multi-characteristic opsin (MCO) gene expression cassette

SUMMARY:
The current study is a non-interventional long-term safety follow-up of the subjects who completed STARLIGHT, in accordance with FDA guidance on recipients of human gene therapy products.

DETAILED DESCRIPTION:
This study is designed to follow subjects with Stargardt Disease (SD) previously enrolled in study NTXMCO-004 (STARLIGHT, NCT05417126). In that study, all 6 enrolled subjects received MCO-010, an ambient light-activated, Multi-Characteristic Opsin (MCO) transgene in an adeno-associated virus serotype 2 (AAV2) vector via intravitreal injection (IVT). MCO-010 has the potential to restore vision irrespective of the underlying gene mutation, and because it is directed at bipolar retinal cells, intact photoreceptors are not required. Further details on MCO-010 and the underlying disease under investigation are included in the protocol for STARLIGHT and are not repeated herein

ELIGIBILITY:
Inclusion Criteria:

* Subjects are eligible to be included in the study only if all of the following criteria apply:

  1. Previously enrolled in study NTXMCO-004 study
  2. Able to comprehend and give informed consent.
  3. Able to comply with testing and all protocol tests.
  4. Agree to participate for the full 4-year study duration to the best of their ability and barring any unforeseen circumstances.

Exclusion Criteria:

* Not applicable. Subjects will be included in this study and will be consented after completion of all assessments at the Week 48 visit for the STARLIGHT study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population eligible to participate will comprise of the 6 subjects previously enrolled in STARLIGHT.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of the long-term safety profile of a single intravitreal injection of MCO-010 | 204 weeks
  Assessment of incidences, nature, and severity of treatment emergent adverse events (TEAEs), serious adverse events (SAEs); intraocular inflammation graded through ocular exam; clinical examination, and intraocular pressure.

SECONDARY OUTCOMES:
Evaluation of the long-term effects on visual acuity of a single intravitreal injection of MCO-010; 1.2E11 gc/eye | 204 weeks
  Change from baseline in BCVA over time in the study eye and fellow eye
Exploration of the long-term impact of MCO-010 on retinal anatomy | 204 weeks
  Assessment of fundus photography and optical coherence tomography (OCT) outcomes over time
Assessment of the long-term durability of MCO-010 induced on gene reporter expression | 204 weeks
  Change from baseline of fundus fluorescence intensity of reporter (mCherry) over time in the study eye and fellow eye

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Samarendra Mohanty, Study Director — Nanoscope Therapeutics Inc.
Locations (2):
- United States (2):
  - Nanocope Clnical Site, Miami, Florida
  - Nanoscope Clinical Site, McAllen, Texas

IPD SHARING:
Plan to Share IPD: Yes
The results of the clinical trial will be made available when the study is completed. The results will be published on this site and be available to conference presentations and publications.
Time Frame: Within a year from the long term monitoring data availability
Access Criteria: IPD sharing access will be subject to data transfer agreement. IPD generated as part of this clinical study may be subject to patient confidentiality.